

## TRIAL STATISTICAL ANALYSIS PLAN

c30563921-01

| BI Trial No.: | 1402-0009 |
|---|---|
| Title: | Relative bioavailability of rosuvastatin (Part 1) and dabigatran (Part 2) given alone and together with BI 1358894 in healthy male subjects (open, single-dose, fixed sequence, two-period crossover design in each trial part) (including Protocol Amendment No.1 [c27867536-02]) |
| Investigational Product: | BI 1358894 |
| Responsible trial statisticians: | |
| | Phone: |
| | Fax: |
| Date of statistical analysis plan: | 21 JAN 2020 SIGNED |
| Version: | 1 |

Proprietary confidential information
© 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

Boehringer Ingelheim
TSAP for BI Trial No: 1402-0009 
Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| 1 | , | ΓΔ | RI | $\mathbf{F}$ | OF · | CO | N | NT | rs |
|---|---|----|----|--------------|--------------|----|---|------|----|
| | • | | | 1 1 | <b>\ / </b> | | | <br> | |

| TITLE PAGE | | |
|---|---|---|
| 1. | TABLE OF CONTENTS | 2 |
| LIST O | TABLES | 4 |
| 2. | LIST OF ABBREVIATIONS | 5 |
| 3. | INTRODUCTION | |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY | |
| <br>5. | ENDPOINTS | |
| 5.<br>5.1 | PRIMARY ENDPOINTS | 9<br>0 |
| 5.1<br>5.2 | SECONDARY ENDPOINTS | |
| 5.2.1 | Key secondary endpoints | |
| 5.2.2 | Secondary endpoints | |
| 5.3.3 | Safety endpoints | 10 |
| | CENTED AL ANALYSIS DEFENDATIONS | 10 |
| 6. | GENERAL ANALYSIS DEFINITIONS | |
| 6.1<br>6.2 | TREATMENTSIMPORTANT PROTOCOL DEVIATIONS | |
| 6.2<br>6.3 | SUBJECT SETS ANALYSED | |
| 0.3 | SUBJECT SETS ANALTSED | 13 |
| 6.5 | POOLING OF CENTRES | 16 |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS | |
| <b>6.7</b> | BASELINE, TIME WINDOWS AND CALCULATED VISITS | 17 |
| 7. | PLANNED ANALYSIS | 18 |
| <b>7.1</b> | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| 7.2 | CONCOMITANT DISEASES AND MEDICATION | 20 |
| 7.3 | TREATMENT COMPLIANCE | <b>20</b> |
| 7.4 | PRIMARY ENDPOINTS | |
| 7.4.1 | Primary analysis of the primary endpoints | 20 |
| 7.4.2.1 | Further exploratory analyses | 21 |
| 7.5 | SECONDARY ENDPOINTS | |
| 7.5.1 | Key secondary endpoints | |
| 7.5.2 | Secondary endpoints | |
| 7.6.2 | Safety endpoints | |
| 7.7 | EXTENT OF EXPOSURE | |
| 7.8 | SAFETY ANALYSIS | 23 |

# **Boehringer Ingelheim**

| T. | ~ | c | 20 |
|------|---|-----|----|
| Page | 3 | OI. | 28 |

| Proprietar | ry confidential information © 2020 Boehringer Ingelheim International Gml | bH or one or more of its affiliated companies |
|---|---|---|
| 7.8.1 | Adverse Events | 23 |
| 7.8.2 | Laboratory data | 24 |
| 7.8.3 | Vital signs | 25 |
| 7.8.4 | ECG | 25 |
| 7.8.5 | Others | 25 |
| 8. | REFERENCES | 26 |
| 10. | HISTORY TABLE | 28 |

Boehringer Ingelheim
TSAP for BI Trial No: 1402-0009
Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## LIST OF TABLES

| Table 6.1: 1 | Treatments and labels used in the analysis | . 12 |
|--------------|--------------------------------------------|------|
| | Subject sets analysed | |
| | History table | |

TSAP for BI Trial No: 1402-0009 

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### LIST OF ABBREVIATIONS 2.

See Medicine Glossary: website: glossary

| Term | Definition / description |
|---|---|
| ALT | Alanine transaminase |
| AST | Aspartate transaminase |
| $\mathrm{AUC}_{0\text{-tz}}$ | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point |
| $\mathrm{AUC}_{0\text{-}\infty}$ | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity |
| BMI | Body mass index |
| BWU | Bioavailability/Bioequivalence, Within-Subject Design, uncontrolled |
| CI | Confidence interval |
| $C_{max}$ | Maximum measured concentration of the analyte in plasma |
| CV | Arithmetic coefficient of variation |
| DILI | Drug induced liver injury |
| gCV | Geometric coefficient of variation |
| gMean | Geometric mean |
| LLT | Lower level term |
| IQRMP | Integrated Quality and Risk Management Plan |
| $\lambda_{\rm z}$ | Terminal rate constant of the analyte in plasma |
| Max | Maximum |
| MedDRA | Medical Dictionary for Regulatory Activities |
| Min | Minimum |
| N | Number non-missing observations |
| P10 | 10th percentile |
| P90 | 90th percentile |
| po | Orally |
| PKS | Pharmacokinetic parameter analysis set |
| Q1 | 1st quartile |
| Q3 | 3rd quartile |
| qd | Once daily |

Boehringer Ingelheim
TSAP for BI Trial No: 1402-0009
Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Term | Definition / description |
|--------|-------------------------------------------|
| R | Reference treatment |
| RAGe | Report Appendix Generator system |
| REP | Residual effect period |
| RPM | Report Planning Meeting |
| SD | Standard deviation |
| SOC | System organ class |
| T | Test treatment |
| TS | Treated set |
| ULN | Upper limit of normal |
| WHO-DD | World Health Organization Drug Dictionary |

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 3. INTRODUCTION

As per ICH E9  $(\underline{1})$ , the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This Trial statistical analysis plan (TSAP) assumes familiarity with the Clinical Trial Protocol (CTP). In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomisation.

Study data (including data entered in the RAVE EDC system and external data provided by suppliers) will be stored in a Clinical Data Repository (CDR).

Pharmacokinetic (PK) and pharmacodynamics (PD) parameters will be calculated using Phoenix WinNonlin TM software (version 6.3 or higher, Certara USA Inc., Princeton, NJ, USA).

The statistical analyses will be performed within the validated working environment CARE, including SAS<sup>TM</sup> (current Version 9.4, by SAS Institute Inc., Cary, NC, USA), and a number of SAS<sup>TM</sup>-based tools (e.g., macros for the analyses of AE data or laboratory data; Report Appendix Generator system (RAGe) for compilation/formatting of the CTR appendices).

## 4. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

All analyses as planned in the CTP will be performed and are described in more detail in this TSAP.

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 5. ENDPOINTS

## 5.1 PRIMARY ENDPOINTS

## **Section 2.1.2 of the CTP:**

*In Part 1 the following pharmacokinetic parameters will be determined for rosuvastatin:* 

- $AUC_{0-\infty}$  (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity)
- $C_{max}$  (maximum measured concentration of the analyte in plasma)

*In Part 2 the following pharmacokinetic parameters will be determined for dabigatran:* 

- $AUC_{0-\infty}$  (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity)
- $C_{max}$  (maximum measured concentration of the analyte in plasma)

## 5.2 SECONDARY ENDPOINTS

## 5.2.1 Key secondary endpoints

This section is not applicable as no key secondary endpoints have been defined in the CTP.

## 5.2.2 Secondary endpoints

## Section 2.1.3 of the CTP:

*In Part 1 the following pharmacokinetic parameter will be determined for rosuvastatin:* 

•  $AUC_{0-tz}$  (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point)

*In Part 2 the following pharmacokinetic parameter will be determined for dabigatran:* 

•  $AUC_{0-tz}$  (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point)

## **5.3.3** Safety endpoints

**Section 2.2.2.4 of the CTP:** *Safety and tolerability of rosuvastatin, dabigatran and BI 1358894 will be assessed based on:* 

- Adverse events (including clinically relevant findings from the physical examination)
- Safety laboratory tests
- 12-lead ECG
- Vital signs (blood pressure, pulse rate)

Boehringer Ingelheim
TSAP for BI Trial No: 1402-0009
Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 6. GENERAL ANALYSIS DEFINITIONS

## 6.1 TREATMENTS

For basic study information on investigational products, assignment of treatment sequences and selection of doses, please see CTP, Sections 3 and 4.

The study consists of 2 trial parts. It is planned that 14 healthy male subjects each will enter either Part 1 or Part 2 of the study. Each part follows a non-randomised, open-label, two-period crossover design with a fixed sequence in healthy male subjects in order to compare the test (T1, T2) and reference (R1, R2) treatments as defined in Table 6.1: 1 below.

Table 6.1: 1 Treatments and labels used in the analysis

| Treati | Short label | |
|---|---|---|
| Part 1 | | |
| R1 | Rosuvastatin, 10 mg tablet, qd | Rosuvastatin |
| T1 | BI 1358894, 2*100 mg tablet + Rosuvastatin, 10 mg tablet, qd | BI+Rosuvastatin |
| Part 2 | | |
| R2 | Dabigatran etexilate, 150 mg capsule, qd | Dabigatran |
| T2 | BI 1358894, 2*100 mg tablet + Dabigatran etex., 150 mg cap, qd | BI+Dabigatran |

**Section 1.2.4 of the CTP:** Based on an effective half-life of 33 h the Residual Effect Period (REP) of BI 1358894 has been determined to be 7 days. The REP for rosuvastatin and dabigatran is approximately 6 and 3 days, respectively. This is the period after the last dose with relevant measurable drug levels and/or pharmacodynamic effects is still likely to be present.

The following separate study phases will be defined for the analyses of adverse events (AEs):

## <u>Part 1:</u>

• **Screening** (ranging from 0:00 h on day of informed consent until first administration time of Rosuvastatin in treatment period 1)

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## • On treatment

- o **Rosuvastatin alone** (labelled "**Rosuvastatin**", including REP; i.e. ranging from the time of first administration of Rosuvastatin in treatment period 1 until 6 days thereafter)
- o **BI+Rosuvastatin** (ranging from time of administration of BI 1358894 + Rosuvastatin in treatment period 2 until 7 days thereafter)
- Follow-up (FU) (labelled "F/U Rosuvastatin", "F/U BI+Rosuvastatin")
  - o F/U Rosuvastatin (ranging from the end of REP of Rosuvastatin in treatment period 1 until the administration of BI+Rosuvastatin in period 2 or until trial termination, whatever occurs first)
  - o **F/U BI+Rosuvastatin** (ranging from the end of REP of BI 1358894 in treatment period 2 until trial termination)

## Part 2:

• Screening (ranging from 0:00 h on day of informed consent until first administration time of Dabigatran in treatment period 1)

## • On treatment

- o **Dabigatran alone** (labelled "**Dabigatran**") (ranging from the time of first administration of Dabigatran in treatment period 1 until 3 days thereafter)
- o **BI+Dabigatran** (ranging from time of administration of BI 1358894 + Dabigatran in treatment period 2 until 7 days thereafter)
- Follow-up (FU) (labelled "F/U Dabigatran", "F/U BI+Dabigatran")
  - o F/U Dabigatran (ranging from the end of REP of Dabigatran in treatment period 1 until the administration of BI+Dabigatran in period 2 or until trial termination, whatever occurs first)
  - o **F/U BI+Dabigatran** (ranging from the end of REP of BI 1358894 in treatment period 2 until trial termination)

**Section 7.3.4 of the CTP:** Note that AEs occurring after the last per protocol contact but entered before final database lock will be reported to Pharmacovigilance only and will not be captured in the trial database.

## The following AE displays will be provided in the report:

Section 15.3 and Appendix 16.1.13.1.8 (for ClinicalTrials.gov and EudraCT only) of the CTR displays:

In these displays, the on-treatment phase will be analysed (labelled with the name of the study treatment (short label)). <u>Screening and Follow up periods will not be included in this analysis</u>.

The following totals will be provided in addition (Section 15.3 only):

- a total over all on treatment phases of study part 1 included in this analysis ("Total Part 1")
- a total over all on treatment phases of study part 2 included in this analysis ("Total Part 2")
- for ClinicalTrials.gov and EudraCT only: a total over all **on treatment phases** included in this analysis ("**Total**")

In Section 15.4 and Appendix 16.2 (Listings) of the CTR displays screening and follow-up periods will be included and no totals will be provided.

Table of vital signs will present results by the above mentioned on treatment phases (Rosuvastatin, BI+Rosuvastatin or Dabigatran, BI+Dabigatran).

For detailed information on the handling of the treatments refer to Technical TSAP ADS (analysis data set) plan and Analysis Data Reviewers guide.

In outputs for ClinicalTrials.gov and EudraCT both study parts will be combined in one table.

## 6.2 IMPORTANT PROTOCOL DEVIATIONS

Data discrepancies and deviations from the CTP will be identified for all treated subjects.

**Section 7.3 of the CTP:** *Important protocol deviation (IPD) categories will be suggested in the IQRM plan, IPDs will be identified no later than in the Report Planning Meeting, and the IPD categories will be updated as needed.* 

Consistency check listings (for identification of deviations of time windows) and a list of protocol deviations (e.g. deviations in drug administration, in blood sampling times, etc.) will be provided to be discussed at the report planning meeting (RPM). At this meeting, all manual deviations identified at the sites by the CRAs and deviations too complex to program will be reviewed by the trial team to decide which are considered important. For definition of important protocol deviations (iPD), and for the process of identification of these, refer to the Boehringer Ingelheim (BI) SOP "Identify and Manage Important Protocol Deviations (iPD)" (2).

If any iPDs are identified, they are to be summarised into categories and will be captured in an accompanying Excel spreadsheet (3). Categories which are considered to be iPDs in this trial are defined in the integrated quality and risk management plan (IQRMP). If the data show other iPDs, the definition in the IQRMP will be supplemented accordingly by the time of the Report Planning Meeting.

The iPDs will be summarised and listed.

## 6.3 SUBJECT SETS ANALYSED

#### Section 7.3 of the CTP:

- Treated set (TS): The treated set includes all subjects who were entered and treated with at least one dose of study drug. The treated set will be used for safety analyses.
- Pharmacokinetic parameter analysis set (PKS): This set includes all subjects in the treated set (TS) who provide at least one PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability (as specified in the following subsection 'Pharmacokinetics'). Thus, a subject will be included in the PKS, even if he contributes only one PK parameter value for one period to the statistical assessment. Descriptive and model based analyses of PK parameters will be based on the PKS. PKS also will be used for the descriptive analyses of PD parameters.

[...]

Plasma concentration data and parameters of a subject will be included in the statistical pharmacokinetic (PK) analyses if they are not flagged for exclusion due to a protocol deviation relevant to the evaluation of PK (to be decided no later than in the Report Planning Meeting) or due to PK non-evaluability (as revealed during data analysis, based on the criteria specified below). Exclusion of a subject's data will be documented in the CTR.

Relevant protocol deviations may be

- Incorrect trial medication taken, i.e. the subject received at least one dose of trial medication the subject was not assigned to
- Incorrect dose of trial medication taken

Plasma concentrations and/or parameters of a subject will be considered as non-evaluable, if for example

- The subject experienced emesis that occurred at or before two times median  $t_{max}$  of the respective treatment (Median  $t_{max}$  is to be determined excluding the subjects experiencing emesis),
- A pre-dose concentration is >5%  $C_{max}$  value of that subject
- Missing samples/concentration data at important phases of PK disposition curve

The descriptive analysis of PK concentrations will be based on the ADS ADPC as described at the beginning of Section 7.

Table 6.3: 1 Subject sets analysed

| | Subj | ject set |
|---------------------------------|------|----------|
| Class of endpoint | TS | PKS |
| Analyses of PK/PD endpoints | | X |
| Safety parameters | X | |
| Demographic/baseline parameters | X | |
| Important protocol deviations | X | |
| Disposition | X | |

## 6.5 POOLING OF CENTRES

This section is not applicable, because the study was performed in only one centre.

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 6.6 HANDLING OF MISSING DATA AND OUTLIERS

Handling of missing data and outliers will be performed as described in the CTP, Section 7.5.

The only exceptions where imputation might be necessary for safety evaluation are AE dates. Missing or incomplete AE dates are imputed according to BI standards (see BI-KMED-BDS-HTG-0035 (4)).

Missing data and outliers of PK/PD data are handled according to BI standards (see 001-MCS-36-472 RD-01) (5).

## 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

The baseline value is defined as the last measurement before trial medication administration in each treatment period.

**Section 6.1 of the CTP:** Exact times of measurements outside the permitted time windows will be documented. The acceptable time windows for screening and the end of trial examination are provided in the CTP Flow Chart.

Study measurements and assessments scheduled to occur 'before' trial medication administration on Day 1 are to be performed and completed within a 3 h-period prior to the trial drug administration.

The acceptable deviation from the scheduled time for vital signs, and laboratory tests will be  $\pm$  60 min.

Starting from a planned time of 48 hours after drug administration (and beyond) a time window of  $\pm$ 120 minutes will be allowed for all procedures.

The acceptable deviations from the scheduled time for PK/PD blood sampling will be:

- $\pm$  15 min for planned times >0:00 and  $\leq$  4 h after trial drug administration
- $\pm$  30 min for planned times > 4h and <48h
- $\pm$  120 min for planned times  $\geq$  48h

The pre-dose sample at planned time -3h is to be drawn within a 3 h-period prior to the trial drug administration.

Adherence to time windows will be checked via the consistency check listings at the RPM.

Unscheduled measurements of laboratory data and vital signs data will be assumed to be repeat measurements of the most recent scheduled measurement (e.g. for follow-up or confirmation of a particular value). Therefore, unscheduled measurements will be assigned to the planned time point of the previous scheduled measurement.

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 7. PLANNED ANALYSIS

If not stated otherwise, the trial parts will be evaluated separately.

Safety analysis (refer to Section 7.8) will be performed by and will be presented in Sections 15.1 to 15.4 of the CTR and in Appendix 16.2 and 16.1.13.1.

Inferential statistical analyses of PK endpoints (refer to Section 7.4 and Section 7.5.2) will also be performed by and will be presented in Section 15.5 of the CTR and in Appendix 16.1.13.3.

Descriptive data analysis of PK/PD endpoints and concentrations will be performed by the at and will be presented in Section 15.6 and Section 15.7 of the CTR.

The format of the listings and tables will follow the BI standards (see BI-KMED-BDS-HTG-0045 (6)) with the exception of those generated for PK-calculations (7).

The individual values of all subjects will be listed, sorted by sequence group, subject number, visit and actual treatment (if appropriate).

The listings will be included in Appendix 16.2 of the CTR.

For end-of-text tables, the set of summary statistics for non-PK parameters is:

N number non-missing observations

Mean arithmetic mean SD standard deviation

Min minimum Median median Max maximum

For analyte concentrations, the following descriptive statistics will additionally be calculated:

CV arithmetic coefficient of variation

gMean geometric mean

gCV geometric coefficient of variation

For PK/PD parameters, the following descriptive statistics will additionally be calculated:

CV arithmetic coefficient of variation

gMean geometric mean

gCV geometric coefficient of variation

P10 10th percentile
Q1 1st quartile
Q3 3rd quartile
P90 90th percentile

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The data format for descriptive statistics of concentrations will be identical to the data format of the respective concentrations. The descriptive statistics of PK parameters will be calculated using the individual values with the number of decimal places as provided by the evaluation program. Then the individual values as well as the descriptive statistics will be reported with three significant digits in the CTR.

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category, as well as the percentage (%). Percentages will be rounded to one decimal place and will be based on all subjects in the respective subject set whether they have non-missing values or not. The category 'missing' will be displayed only if there are actually missing values.

Units of variables should be given in the titles or column/row descriptors in square brackets (e.g. [mg]).

## Exclusion of PK parameters

The ADS ADPP (PK parameters) contains column variables indicating inclusion/exclusion (APEXC) of a PK parameter and an analysis flag comment (APEXCO). All analyses based on the PKS will include parameters if they are not flagged for exclusion, that is APEXC is equal to "Included".

## Exclusion of PK concentrations

The ADS ADPC (PK concentrations per time-point or per time-interval) contains column variables ACEXC and ACEXCO indicating inclusion/exclusion (ACEXC) of a concentration and an analysis flag comment (ACEXCO). Exclusion of a concentration depends on the analysis flag comment ACEXCO. For example, if ACEXCO is set to 'ALL CALC', the value will be excluded for all types of analyses based on concentrations. If ACEXCO is set to 'DESC STATS' the value will be excluded from descriptive evaluations per planned time point/time interval. If ACEXCO contains the addition 'TIME VIOLATION' or 'TIME DEVIATION' the value can be used for further analyses based on actual times. If ACEXCO is set to 'HALF LIFE', the value will be excluded from half-life calculation (and, as a consequence, any calculation that relies on  $\lambda_z$ ) only; the value is included for all other analyses.

Further details are given in 001-MCS-36-472\_RD-01 "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies" (5) and 001-MCS-36-472\_RD-03 "Description of Analytical Transfer Files and PK/PD Data Files" (11).

## 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the report, based on the TS.

The data will be summarised in total, separately for trial part 1 and part 2.

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 7.2 CONCOMITANT DISEASES AND MEDICATION

Frequency tables are planned for this section of the report, based on the TS.

Concomitant diseases will be coded using the coding system of the Medical Dictionary for Drug Regulatory Activities (MedDRA). Medications will be coded using the World Health Organization Drug Dictionary (WHO-DD). The coding version number will be displayed as a footnote in the respective output.

The diagnoses and medications will be listed. Subjects without any concomitant diagnoses or concomitant therapies should be marked with a "No" in the respective column.

The relevance of the concomitant therapies to the evaluation of PK will be decided no later than at the RPM.

## 7.3 TREATMENT COMPLIANCE

**Section 4.3 of the CTP:** Compliance will be assured by administration of all trial medication in the study centre under supervision of the investigating physician or a designee. The measured plasma concentrations of trial medication will provide additional confirmation of compliance.

It is not intended to list the compliance separately. Any deviations from complete intake will be addressed in the RPM (cf. TSAP <u>Section 6.2</u>) and described in the CTR.

## 7.4 PRIMARY ENDPOINTS

Relative bioavailability of rosuvastation (part 1) and dabigatran (part 2) is to be determined on the basis of the primary endpoints  $AUC_{0-\infty}$ ,  $C_{max}$  (see Section 5.1).

## 7.4.1 Primary analysis of the primary endpoints

**Section 7.3.1 of the CTP:** The statistical model used for the analysis of the primary endpoints will be an analysis of variance (ANOVA) model on the logarithmic scale. That is, the PK endpoints will be log-transformed (natural logarithm) prior to fitting the ANOVA model. This model will include effects accounting for the following sources of variation: subjects and treatment. The effect 'subjects' will be considered as random, whereas 'treatment' will be considered as fixed. The model is described by the following equation:

$$y_{km} = \mu + s_m + \tau_k + e_{km}$$
, where

- $y_{km} = logarithm \ of \ response \ measured \ on \ subject \ m \ receiving \ treatment \ k,$
- $\mu = the overall mean$ ,

TSAP for BI Trial No: 1402-0009 Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- $s_m$  = the effect associated with the  $m^{th}$  subject, m = 1, 2, ..., n
- $\tau_k = the \ k^{th} \ treatment \ effect, \ k = 1, 2,$
- $e_{km}$  = the random error associated with the  $m^{th}$  subject who received treatment k.

where  $s_m \sim N(0, \sigma_w^2)$  i. i. d.,  $e_{km} \sim N(0, \sigma_w^2)$  i.i.d. and  $s_m$ ,  $e_{km}$  are independent random variables.

Point estimates for the ratios of the geometric means (test/reference) for the primary endpoints (see Section 2.1) and their two-sided 90% confidence intervals (CIs) will be provided.

For each endpoint, the difference between the expected means for log(T)-log(R) will be estimated by the difference in the corresponding adjusted means (Least Squares Means). Additionally their two-sided 90% confidence intervals will be calculated based on the residual error from the ANOVA and quantiles from the t-distribution. These quantities will then be back-transformed to the original scale to provide the point estimate and 90% CIs for each endpoint.

The implementation for this analysis will be accomplished by using the CSD macros. The following SAS code can be used:

```
PROC MIXED DATA=indata;
```

CLASS subject treatment;

MODEL logkp = treatment / HTYPE = 2 SOLUTION CL alpha=0.1;

RANDOM subject;

LSMEANS treatment /CL alpha=(1-&CONFLEV/100) pdiff=control("Ref trt");

RUN;

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 7.5 SECONDARY ENDPOINTS

## 7.5.1 Key secondary endpoints

This section is not applicable as no key secondary endpoint has been specified in the protocol.

## 7.5.2 Secondary endpoints

The secondary PK parameter  $AUC_{0-tz}$  for rosuvastatin (part 1) and dabigatran (part 2) will be assessed using the same methods as described for the primary endpoints.

## 7.6.2 Safety endpoints

Refer to TSAP <u>Section 7.8</u> for a description of the analysis of safety and tolerability of BI 1358894.

## 7.7 EXTENT OF EXPOSURE

Descriptive statistics are planned for this section of the report based on the TS. The date and time of drug administration will be listed for each subject.

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the TS.

The safety data for treated subjects who failed to complete the study (dropouts or withdrawals) will be reported as far as their data are available. All withdrawals will be documented and the reason for withdrawal recorded.

## 7.8.1 Adverse Events

AEs will be coded with the most recent version of MedDRA.

The analyses of AEs will be descriptive in nature and will be based on BI standards as presented in "Analysis and Presentation of Adverse Event Data from Clinical Trials – Display Template" [BI-KMED-BDS-HTG-0041] (8). All analyses of AEs will be based on the number of subjects with AEs and not on the number of AEs.

For analysis multiple AE occurrence data on the eCRF will be collapsed into one AE provided that all of the following applies:

- All AE attributes are identical (lower level term (LLT), intensity, action taken, therapy required, seriousness, reason for seriousness, relationship, outcome, AE of special interest (AESI))
- The occurrences were time-overlapping or time-adjacent (time-adjacency of two occurrences is given if the second occurrence started within one hour after end of the first occurrence).

The analysis of AEs will be based on the concept of treatment emergent AEs. That means that all AEs will be assigned to screening or on-treatment phases as defined in Section 6.1. AEs will be analysed based on actual treatments, as defined in Table 6.1: 1

## **Section 5.2.6.1.4 of the CTP:** *The following are considered as AESIs:*

- *Hepatic injury* 
  - A hepatic injury is defined by the following alterations of hepatic laboratory parameters:
    - An elevation of AST (aspartate transaminase) and/or ALT (alanine transaminase) ≥3-fold ULN combined with an elevation of total bilirubin ≥2-fold ULN measured in the same blood sample, or
    - Aminotransferase (ALT, and/or AST) elevations  $\geq$ 10 fold ULN

These lab findings constitute a hepatic injury alert and the subjects showing these lab abnormalities need to be followed up according to the 'DILI checklist' provided in the ISF. In case of clinical symptoms of hepatic injury (icterus, unexplained encephalopathy, unexplained coagulopathy, right upper quadrant abdominal pain,

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

etc.) without lab results (ALT, AST, total bilirubin) available, the Investigator should make sure that these parameters are analysed, if necessary in an unscheduled blood test. Should the results meet the criteria of hepatic injury alert, the procedures described in the DILI checklist should be followed.

According to ICH E3 (9), AEs classified as 'other significant' need to be reported and will include those non-serious and non-significant AE with

- (i) 'action taken = discontinuation' or 'action taken = reduced', or
- (ii) marked haematological and other lab abnormalities or lead to significant concomitant therapy as identified by the Clinical Monitor/Investigator at a RPM.

An overall summary of AEs (including AESIs and other significant AEs) will be presented.

The frequency of subjects with AEs will be summarised by treatment, primary system organ class (SOC) and preferred term (PT). Separate tables will be provided for subjects with other significant AEs according to ICH E3 (2), for subjects with serious AEs, for subjects with drug-related AEs, for subjects with drug related serious adverse events and for subjects with AESIs. In addition, the frequency of subjects with AEs will be summarised by treatment, worst intensity, primary system organ class (SOC) and preferred term (PT). The SOCs and PTs will be sorted by frequency (within SOC). The MedDRA version number will be displayed as a footnote in the respective output.

In addition, frequencies of subjects with non-serious AEs that had an incidence of > 5% for at least one treatment will be summarised by treatment, primary SOC and PT.

For disclosure of adverse events on EudraCT, additional information not included in a standard AE analysis will be performed. The following three entries will be created:

- Adverse Events per arm for disclosure on EudraCT
- Non-serious Adverse Events for disclosure on EudraCT
- Serious Adverse Events for disclosure on EudraCT

## 7.8.2 Laboratory data

The analyses of laboratory data will be descriptive in nature and will be based on BI standards [BI-KMED-BDS-HTG-0042] (10).

Laboratory data will be analysed qualitatively via comparison of laboratory data to their reference ranges. Values outside the reference range as well as values defined as possibly clinically significant will be flagged in the data listings.

Clinically relevant findings in laboratory data will be reported as baseline conditions (at screening) or as AEs (during the trial) if judged clinically relevant by the investigator, and will be analysed as such.

It is the investigator's responsibility to decide whether a lab value is clinically significantly abnormal or not (at the RPM/DBLM at the latest).

Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Descriptive statistics of laboratory data including change from baseline (=screening) will be calculated by planned time point based on the worst value of the subject at that planned time point (or assigned to that planned time point).

## 7.8.3 Vital signs

For vital signs (blood pressure and pulse rate), descriptive statistics including change from baseline will be calculated by planned time point based on the last value of the subject at that planned time point (or assigned to that planned time point). In the listing the difference from baseline will also be displayed.

Clinically relevant findings in vital signs will be reported as AEs.

## **7.8.4** ECG

ECG recordings will be checked by the investigator for pathological results. Clinically relevant abnormal findings for ECG will be listed under 'Relevant Medical History / Baseline Conditions' (if they pre-exist prior to trial inclusion) or will be reported as AEs (if they occurred during treatment), and will be analysed as such.

## **7.8.5** Others

## Physical examination

Physical examination findings will be reported as relevant medical history/baseline condition (i.e., a condition already existent before intake of study drug) or as AE and will be summarised as such. No separate listing or analysis of physical examination findings will be prepared.

#### REFERENCES 8.

| 1. | CPMP/ICH/363/96: "Statistical Principles for Clinical Trials", ICH Guideline Topic E9, Note For Guidance on Statistical Principles for Clinical Trials, current version. |
|---|---|
| 2. | 001-MCS-40-413: "Identify and Manage Important Protocol Deviations (iPD) ", current version, IDEA for CON. |
| 3. | BI-KMED-COPS-TMP-0001: "iPD log", current version; KMED. |
| 4. | <i>BI-KMED-BDS-HTG-0035</i> : "Handling of Missing and Incomplete AE Dates", current version; KMED. |
| 5. | 001-MCS-36-472_RD-01: "Noncompartmental Pharmacokinetic/Pharmacodynamic Analyses of Clinical Studies", current version; IDEA for CON. |
| 6. | <i>BI-KMED-BDS-HTG-0045</i> : "Standards for Reporting of Clinical Trials and Project Summaries", current version; KMED. |
| 7. | 001-MCS-36-472: "Standards and processes for analyses performed within Clinical Pharmacokinetics/Pharmacodynamics", current version; IDEA for CON. |
| 8. | <i>BI-KMED-BDS-HTG-0041</i> : "Analysis and Presentation of Adverse Event Data from Clinical Trials – Display Template", current version; KMED. |
| 9. | CPMP/ICH/137/95: "Structure and Content of Clinical Study Reports", ICH Guideline Topic E3; Note For Guidance on Structure and Content of Clinical Study Reports, current version. |
| 10. | BI-KMED-BDS-HTG-0042: "Handling, Display and Analysis of Laboratory Data", current version; KMED. |
| 11. | 001-MCS-36-472_RD-03: "Description of Analytical Transfer Files and PK/PD Data Files", current version; IDEA for CON. |

Boehringer Ingelheim
TSAP for BI Trial No: 1402-0009
Proprietary confidential information © 2020 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **HISTORY TABLE 10.**

Table 10: 1 History table

| Version | Date | Author | Sections | Brief description of change |
|---------|-------------|--------|----------|-----------------------------|
| | (DD-MMM-YY) | | changed | |
| 1 | 21-JAN-2020 | | None | This is the final TSAP. |